CLINICAL TRIAL: NCT04865237
Title: A Dose Finding Human Experimental Infection Study in Healthy Subjects Using a GMP-produced SARS-COV-2 Wild Type Strain
Brief Title: SARS-CoV-2 Human Challenge Characterisation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Hvivo (Industry); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20IC6437
Record Dates: First submitted 2021-04-01; First posted 2021-04-29 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Covid19; SARS-CoV Infection; Corona Virus Infection; Coronavirus; COVID-19
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — remdesivir

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers Dose Level 1 (Experimental): Dose Level 1: SARS-CoV-2, intranasally (10^1 TCID50 dose)
  Interventions: Biological: SARS-CoV-2 Virus 1x10^1 TCID50; Drug: Remdesivir
- Healthy Volunteers Dose Level 2 (Experimental): Dose Level 2: SARS-CoV-2, intranasally (10^2 TCID50 dose)
  Interventions: Drug: Remdesivir; Biological: SARS-CoV-2 Virus 1x10^2 TCID50
- Healthy Volunteers Dose Level 3 (Experimental): Dose Level 3: SARS-CoV-2, intranasally (10^3 TCID50 dose)
  Interventions: Drug: Remdesivir; Biological: SARS-CoV-2 Virus 1x10^3 TCID50

INTERVENTIONS:
Biological: SARS-CoV-2 Virus 1x10^1 TCID50 — SARS-CoV-2, intranasally, (1x10^1 TCID50)
  Arms: Healthy Volunteers Dose Level 1
Drug: Remdesivir — VEKLURY™
  Other Names: VEKLURY™
Biological: SARS-CoV-2 Virus 1x10^2 TCID50 — SARS-CoV-2, intranasally, (1x10^2 TCID50)
  Arms: Healthy Volunteers Dose Level 2
Biological: SARS-CoV-2 Virus 1x10^3 TCID50 — SARS-CoV-2, intranasally, (1x10^3 TCID50)
  Arms: Healthy Volunteers Dose Level 3

SUMMARY:
This is a dose optimisation study in healthy adults aged 18-30 who will be experimentally inoculated with SARS-CoV-2. The aim is to cause PCR-confirmed upper respiratory infection in the majority of challenged individuals with minimal or no illness, providing data on the course of COVID-19 and the immune response to SARS-CoV-2 infection. This will establish an optimised dose and study design that will then be used to evaluate the efficacy of treatment and vaccine candidates plus level and duration of immune protection in follow-on trials.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the Investigator.
2. Male or female, age between 18 and 30 years inclusive (at the time of consent)
3. Seronegative to the challenge virus SARS-CoV-2, no history of SARS-CoV-2 infection and no previous participation in a SARS-CoV-2 vaccine trial.
4. Female participants with a documented menstrual period within 28 days before the inoculation (unless using a contraceptive method that suppressed menstruation as indicated in the study protocol) and willing and able to use contraception as described in the study protocol from 2 weeks before the scheduled date of viral challenge until 90 days after receipt of the final dose of rescue medication. Negative urine pregnancy tests will be required at screening and on day 0 prior to inoculation. On admission to the quarantine unit a Negative serum beta human chorionic gonadotropin (β-hCG) is required.

Contraceptive requirements:

Established use of hormonal methods of contraception described below (for 2 weeks prior to the first study visit). When hormonal methods of contraception are used, male partners are required to use a condom with a spermicide:

1. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: i. oral ii. intravaginal iii. transdermal
2. . progestogen-only hormonal contraception associated with inhibition of ovulation: i. oral ii. injectable iii. implantable
3. Intrauterine device (IUD)
4. . Intrauterine hormone-releasing system (IUS)
5. . Bilateral tubal ligation
6. . Male sterilisation (with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate) where the vasectomised male is the sole partner for that woman.
7. . True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

5 Men who are willing to use one of the contraception methods described in the study protocol, from the time of the date of viral challenge, until 90 days after receipt of the final dose of study medication.

Contraceptive requirements:

1. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the study virus or Remdesivir.
2. Male sterilisation with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study.
3. In addition, for female partners of child bearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female subjects.
4. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

   In addition to the contraceptive requirements above, male subjects must agree not to donate sperm following discharge from quarantine until 90 days after the date of study virus or Remdesivir. (whichever occurs last).

   6 In good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with subject safety, as defined by medical history, physical examination and routine laboratory tests, ECG, and Chest X-Ray and determined by the Investigator at an admission evaluation.

   7 Subjects will have a documented medical history either prior to entering the study and/or following medical history review with the study physician at screening 8 Using the QCOVID tool, an absolute risk of COVID-associated death of 1 in 250,000 (0.0004%) or less and COVID-associated hospital admission of 1 in 5000 (0.02%) or less, unless deemed unnecessary by the CI and PI with advice from the DSMB following a formal interim assessment (see below) 9 Willing and able to commit to participation in the study

   Exclusion Criteria:

   Any potential subject who meet any of the criteria below will be excluded from participating in this study.

   Clinical history
   1. History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory, dermatological, gastrointestinal, endocrine, haematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological, psychiatric illness. Specifically:

      1. Subjects with any history of physician diagnosed and/or objective test confirmed asthma, chronic obstructive pulmonary disease, pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology or who have experienced:

         * Significant/severe wheeze in the past
         * Respiratory symptoms including wheeze which has ever resulted in hospitalisation
         * Known bronchial hyperreactivity to viruses
      2. History of thromboembolic, cardiovascular or cerebrovascular disease
      3. History or evidence of diabetes mellitus
      4. Any concurrent serious illness including history of malignancy that could interfere with the aims of the study or a subject completing the study. Basal cell carcinoma within 5 years of treatment or with evidence of recurrence is also an exclusion
      5. Migraine with associated neurological symptoms such as hemiplegia or vision loss. Cluster headache/migraine or prophylactic treatment for migraine
      6. History or evidence of autoimmune disease or known immunodeficiency of any cause.
      7. Other major disease that, in the opinion of the Investigator, could interfere with a subject completing the study and necessary investigations.
      8. Immunosuppression of any type
   2. Any significant abnormality altering the anatomy or function of the nose or nasopharynx in a substantial way (including loss of or alterations in smell or taste), a clinically significant history of epistaxis (large nosebleeds) within the last 3 months, nasal or sinus surgery within 6 months of inoculation.
   3. Clinically active rhinitis (including hay fever) or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine.
   4. History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the PI.
   5. History or presence of alcohol addiction, or excessive use of alcohol (average weekly intake in excess of 28 units alcohol; one unit being a half glass of beer, a small glass of wine or a measure of spirits), or use of drugs of abuse
   6. Psychiatric illness including subjects with a history of depression and/or anxiety with associated severe psychiatric comorbidities, for example psychosis. Specifically,

      1. Subjects with history of anxiety-related symptoms of any severity within the last 2 years if the Generalized Anxiety Disorder-7 score is ≥4
      2. Subjects with a history of depression of any severity within the last 2 years if the Patient Health Questionnaire-9 score is ≥4
   7. Subjects who have smoked ≥5 pack years at any time [5 pack years is equivalent to one pack of 20 cigarettes a day for 5 years]).

      • Subjects who have smoked <5 pack years - at any time in the 3 months prior to admission to the quarantine unit they have used tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) or electronic cigarettes.
   8. Family history of 1st degree relative aged 50 years or less with sudden cardiac or unexplained death
   9. Family History of Severe COVID or response to any other viral disease e.g. Guillain-Barré Measurements and investigations
   10. A total body weight of ≤ 50kg and a Body Mass Index (BMI) ≤18 kg/m2 and ≥28 kg/m2. The upper limit of BMI may be increased to ≤ 30kg/m2 at the PI's discretion, in the case of physically fit muscular individual
   11. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
   12. Any clinically significant abnormal finding on screening biochemistry, haematology and microbiology blood tests or urinalysis i.e. grade 1 lab abnormalities (or above, see Appendix 3 Toxicity Grading Scale for Laboratory AEs) apart from minor deviations which are clinically acceptable and approved by the Principal Investigator

       1. Elevated random glucose and HbA1C
       2. Positive HIV, active/chronic hepatitis A, B or C test.
       3. Confirmed positive test for drugs of abuse on admission and urinary cotinine at quarantine.
   13. A forced expiratory volume in 1 second (FEV1) and a forced vital capacity (FVC) <80% of predicted value calculated using ATS/ERS guidance (refer to section 5, respiratory samples)
   14. Twelve-lead ECG recording with clinically relevant abnormalities as judged by the study physician/PI.
   15. Echocardiogram outside normal parameters at baseline Recent respiratory infection
   16. History of, or currently active symptoms suggestive of upper or lower respiratory tract infection (including reduced sense of taste and smell, raised body temperature and/or persistent cough) within 6 weeks prior to viral challenge.
   17. Presence of cold-like symptoms and/or fever (defined as subject presenting with a temperature reading of >37.9ºC) on Day -2, Day -1 and/or pre-challenge on Day 0.
   18. Evidence of any respiratory viruses (on nasopharyngeal swab analysis) prior to challenge virus inoculation on admission to the quarantine unit. These include:

       VIRUSES:
       * Adenovirus
       * Coronavirus HKU1
       * Coronavirus NL63
       * Coronavirus 229E
       * Coronavirus OC43
       * Human Metapneumovirus
       * Human Rhinovirus/Enterovirus
       * Influenza A
       * Influenza A/H1
       * Influenza A/H3
       * Influenza A/H1-2009
       * Influenza B
       * Parainfluenza Virus 1
       * Parainfluenza Virus 2
       * Parainfluenza Virus 3
       * Parainfluenza Virus 4
       * Respiratory Syncytial Virus

       BACTERIA:
       * Bordetella parapertussis
       * Bordetella pertussis
       * Chlamydia pneumoniae
       * Mycoplasma pneumoniae Receipt of medications and interventions
   19. Evidence of a live vaccine within 60 days prior to the planned date of viral challenge, a non-live vaccine within 30 days prior to the planned date of viral challenge, or intention to receive any vaccination(s) before the day 28 follow-up visit. (NB. No travel restrictions applied after the Day 28 Follow-up visit).
   20. Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned date of viral challenge or planned during the 3 months after the final visit.
   21. Medications

       1. Use of any medication or product (prescription or over-the-counter), for symptoms of hayfever, nasal congestion or respiratory tract infections or dermatitis/eczema including the use of regular nasal or medium-high potency dermal corticosteroids, antibiotics and First Defence™ (or generic equivalents) within 7 days prior to the planned date of viral challenge apart from those described and allowed in Permitted Medication or agreed by the Principle Investigator
       2. Receipt of any investigational drug within 3 months prior to the planned date of viral challenge.
       3. Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge.
       4. Prior inoculation with a virus from the same virus-family as the challenge virus.
       5. Receipt of systemic (intravenous and/or oral) glucocorticoids or systemic antiviral drugs within 6 months prior to the planned date of viral challenge.
       6. Over the counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date of viral challenge had exceeded the maximum permissible 24-hour dose (e.g., >4g per day of paracetamol over the preceding week).
       7. Use or anticipated use within 7 days prior to the planned date of viral challenge and during the conduct of the study of concomitant medications (prescription and/or non-prescription), including vitamins or herbal and dietary supplements within the specified windows.
       8. Chronically used medications, vitamins or dietary supplements, including any medication known to be a moderate/potent inducer or inhibitor of cytochrome P450 enzymes, within 21 days prior to the planned date of viral challenge.
       9. Subjects who have received any systemic chemotherapy agent, immunoglobulins, or other cytotoxic or immunosuppressive drugs at any time.
   22. Prior participation in another human viral challenge study in the preceding 12 months taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.
   23. Any nasal sampling procedure in the 6 months before date of expected viral challenge in this study (excluding study tolerance test or routine tests for COVID-19) General
   24. Subject was mentally or legally incapacitated in the opinion of the Investigator.
   25. Females who:

       1. Are breastfeeding within 6 months of study commencement, or
       2. Had been pregnant within 6 months prior to the study, or
       3. Had a positive pregnancy test at any point during screening or prior to inoculation with challenge virus
   26. Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 2 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease Other
   27. Was employed or was a first-degree relative of anyone employed by the Sponsor, a participating clinical trial site, or any Contract Research Organisation involved in the study.
   28. Any other reason that the Investigator considered made the subject unsuitable to participate.
   29. Participants with no knowledge of their family history

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - hVIVO Services Ltd, QMB Bioenterprise building, London
  - Royal Free Foundation Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou J, Singanayagam A, Goonawardane N, Moshe M, Sweeney FP, Sukhova K, Killingley B, Kalinova M, Mann AJ, Catchpole AP, Barer MR, Ferguson NM, Chiu C, Barclay WS. Viral emissions into the air and environment after SARS-CoV-2 human challenge: a phase 1, open label, first-in-human study. Lancet Microbe. 2023 Aug;4(8):e579-e590. doi: 10.1016/S2666-5247(23)00101-5. Epub 2023 Jun 9. PMID 37307844
- [Derived] Wagstaffe HR, Thwaites RS, Sidhu JK, Lindeboom RGH, Kretschmer L, Worlock KB, Dratva LM, Huang A, Ascough S, Papargyris L, McKendry R, Collins AM, Xu J, Lemm NM, Killingley B, Kalinova M, Mann A, Catchpole A, Swadling L, Tsang JS, Maini MK, Noursadeghi M, Nikolic MZ, Teichmann SA, Openshaw PJM, Chiu C. Pre-existing and early cellular immune factors correlate with functionally complete protection against primary controlled human SARS-CoV-2 infection. Nat Commun. 2025 Dec 7;17(1):312. doi: 10.1038/s41467-025-67017-8. PMID 41354730
- [Derived] Trender W, Hellyer PJ, Killingley B, Kalinova M, Mann AJ, Catchpole AP, Menon D, Needham E, Thwaites R, Chiu C, Scott G, Hampshire A. Changes in memory and cognition during the SARS-CoV-2 human challenge study. EClinicalMedicine. 2024 Sep 21;76:102842. doi: 10.1016/j.eclinm.2024.102842. eCollection 2024 Oct. PMID 39364271
- [Derived] Killingley B, Mann AJ, Kalinova M, Boyers A, Goonawardane N, Zhou J, Lindsell K, Hare SS, Brown J, Frise R, Smith E, Hopkins C, Noulin N, Londt B, Wilkinson T, Harden S, McShane H, Baillet M, Gilbert A, Jacobs M, Charman C, Mande P, Nguyen-Van-Tam JS, Semple MG, Read RC, Ferguson NM, Openshaw PJ, Rapeport G, Barclay WS, Catchpole AP, Chiu C. Safety, tolerability and viral kinetics during SARS-CoV-2 human challenge in young adults. Nat Med. 2022 May;28(5):1031-1041. doi: 10.1038/s41591-022-01780-9. Epub 2022 Mar 31. PMID 35361992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study met the primary outcome of a 50% infection rate in the first, lowest dose group. Therefore, there was no further enrolment into the higher dose level groups (Dose Level 2 or 3).
Groups:
- Healthy Volunteers Dose Level 1: Healthy volunteers given SARS-CoV-2 virus at 10^1 TCID50 dose +/- Remdesivir: VEKLURY™
- Healthy Volunteers Dose Level 2: Healthy volunteers given SARS-CoV-2 virus at 10^2 TCID50 dose +/- Remdesivir: VEKLURY™
- Healthy Volunteers Dose Level 3: Healthy volunteers given SARS-CoV-2 virus at 10^3 TCID50 dose +/- Remdesivir: VEKLURY™
Period: Overall Study
Arm/Group | Healthy Volunteers Dose Level 1 | Healthy Volunteers Dose Level 2 | Healthy Volunteers Dose Level 3
Started | 36 | 0 | 0
Completed | 36 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy Volunteers Dose Level 1
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (2.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Unsolicited Adverse Events in Healthy Participants Challenged With Wild Type SARS-CoV-2
Description: To evaluate the safety of wild type SARS-CoV-2 challenge in healthy participants by assessing occurrence of unsolicited AEs within 30 days post-viral challenge (Day 0) up to Day 28 follow up.
Time Frame: Day 0 to 28 (28 days)
Population: All subjects
Measure: Number; unit: Unsolicited Adverse Events
Groups:
- Healthy Volunteers Dose Level 1: Healthy volunteers given SARS-CoV-2 virus at 10^1 TCID50 +/- Remdesivir: VEKLURY™
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Unsolicited Adverse Events | 45

2. Primary Outcome: Number of SAEs Related to Viral Challenge
Description: To evaluate the safety of wild type SARS-CoV-2 challenge in healthy participants by assessing occurrence of SAEs related to the viral challenge from the viral challenge (Day 0) up to Day 28 follow up.
Time Frame: Day 0 to 28 (28 days)
Population: Healthy volunteers given SARS-CoV-2 virus at 10^1 TCID50 +/- Remdesivir: VEKLURY™
Measure: Number; unit: SAE events
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
SAE events | 0

3. Primary Outcome: Number of Participants With Laboratory Confirmed Infections
Description: To identify a SARS-Cov-2 inoculum dose that safely induces laboratory confirmed infection in ≥50% of participants (ideally between 50% and 70%). Laboratory confirmed infection is defined as two quantifiable greater than lower limit of quantification (≥LLOQ) RT-PCR measurements from mid turbinate and/or throat samples, reported on 2 or more consecutive timepoints, starting from 24 hours post-inoculation and up to discharge from quarantine.
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Population: 36 individuals were challenge but two were excluded from the analysis due to sero-conversion prior to the viral challenge.
Measure: Number; unit: infected participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 34
infected participants | 18

4. Secondary Outcome: Number of Patients With Laboratory Confirmed Infections by Mid-turbinate and/or Throat Swabs
Description: To further assess SARS-CoV-2 viral infection rates in upper respiratory samples in healthy volunteers, by inoculum dose.
  To assess the incidence of laboratory confirmed infection rates using a) mid turbinate samples, b) throat swabs, and c) both mid turbinate and throat swabs, as defined by:
  * Variant 2: Occurrence of at least two quantifiable (≥LLOQ) RT-PCR measurements, reported on 2 or more consecutive timepoints, starting from 24 hours post-inoculation and up to discharge from quarantine.
  * Variant 3: Occurrence of at least two detectable (≥LLOD) RT-PCR measurements, reported on 2 or more consecutive timepoints, starting from 24 hours post-inoculation and up to discharge from quarantine.
  * Variant 4: Occurrence of at least one quantifiable (≥LLOQ) SARS-CoV-2 viral cell culture measurement, starting from 24 hours post-inoculation and up to discharge from quarantine.
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Measure: Number; unit: infected participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 34
infected participants | 18

5. Secondary Outcome: Number of Symptomatic SARS-Cov-2 Infected Participants
Description: To assess the incidence of symptomatic SARS-CoV-2 infection, in healthy volunteers, by inoculum dose To assess the incidence of lab-confirmed symptomatic SARS-CoV-2 infection using a) mid turbinate samples, b) throat swabs, and c) both mid turbinate and throat swabs,
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Population: Of the 34, participants, 18 participants had confirmed SARS-CoV-2 infections.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 18
Participants | 14

6. Secondary Outcome: SARS-CoV-2 Viral Dynamics (VL-AUC) in Upper Respiratory Samples in Healthy Volunteers
Description: To assess the viral dynamics using a) mid turbinate samples, and b) throat swabs as measured by the area under the viral load-time curve (VL-AUC) of SARS-CoV-2 as determined by qRT-PCR, starting from 24 hours post-inoculation and up to discharge from quarantine.
Time Frame: From 24 hours post-inoculation to 312 hours post-inoculation
Measure: Mean (Standard Deviation); unit: hours*Log10 FFU/mL
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
hours*Log10 FFU/mL | 171.154 (193.2885)

7. Secondary Outcome: SARS-CoV-2 Induced Symptoms in Healthy Volunteers by the Mean Sum Total Symptom Score
Description: Sum total symptoms diary card score: sum total clinical symptoms (TSS) as measured by graded symptom scoring system, starting one day post-viral challenge (Day 1) up to discharge from quarantine. Symptoms are graded on a scale from 0 (no symptoms) to 3 (bothersome symptoms impacting involvement in activities). The sum total symptom score was based on the symptom diary cards that were filled out 3 times per day from the first (morning) assessment on Day 1 until the first (morning) assessment on Day 14 (planned day of quarantine discharge). Each assessment consisted of the grades given by the subjects to a list of 19 symptoms on the symptom diary card. Individual total symptom scores were derived for each assessment as the total of all of the grades given on the individual diary card. This could range from 0 (if all symptoms graded as 0) to 59 (if all symptoms graded as 3 and shortness of breath and wheeze were graded as 4).
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Measure: Mean (Standard Deviation); unit: Sum Total Symptom Score
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Sum Total Symptom Score | 26.8 (42.25)

8. Secondary Outcome: Number of Participants With Incidence of SARS-CoV-2 Illness in Healthy Volunteers
Description: The incidence of:
  * Upper Respiratory Tract illness (URT)
  * Lower Respiratory Tract illness (LRT)
  * Systemic illness (SI)
  * Febrile illness (FI)
  * Proportion of Subjects with Grade 3 symptoms on any occasion at any time from the last assessment on Day 0 to quarantine discharge
  * Proportion of Subjects with Grade 2 or higher symptoms on any occasion at any time from the last assessment on Day 0 to quarantine discharge
  * Proportion of Subjects with Grade 2 or higher Symptoms on two separate occasions at any time from the last assessment on Day 0 to quarantine discharge
  * Proportion of Subjects with any symptom (grade >=1) on any occasion at any time from the last assessment on Day 0 to quarantine discharge
  * Proportion of Subjects with any symptom (grade >=1) on two separate occasions at any time from the last assessment on Day 0 to quarantine discharge
Time Frame: Day 0 to discharge from Quarantine, up to a maximum of 17 days
Measure: Number; unit: participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
participants | 20

9. Secondary Outcome: SARS-CoV-2 Viral Dynamics (Peak Viral Load) in Upper Respiratory Samples in Healthy Volunteers
Description: To assess the viral dynamics using a) mid turbinate samples, and b) throat swabs as measured by peak viral load of SARS-CoV-2 as defined by the maximum viral load determined by quantifiable (≥LLOQ) qRT-PCR measurements, starting from 24 hours post-inoculation and up to discharge from quarantine.
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
log10 copies/mL | 4.5764 (4.50600)

10. Secondary Outcome: SARS-CoV-2 Viral Dynamics (Duration) in Upper Respiratory Samples in Healthy Volunteers
Description: To assess the viral dynamics using a) mid turbinate samples, and b) throat swabs as measured by duration of SARS-CoV-2 quantifiable (≥LLOQ) qRT-PCR measurements, starting from 24 hours post-inoculation and up to discharge from quarantine. Duration is defined as the time (hours) from the first quantifiable of the two viral quantifiable positives used to assess infection until first confirmed undetectable assessment after their peak measure (after which no further virus is detected).
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Measure: Median (Inter-Quartile Range); unit: Duration in Days (Mid-Turbinate)
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Duration in Days (Mid-Turbinate) | 12.52 [11.50 to 14.50]

11. Secondary Outcome: SARS-CoV-2 Viral Dynamics (Incubation Period) in Upper Respiratory Samples in Healthy Volunteers
Description: To assess the viral dynamics using a) mid turbinate samples, and b) throat swabs as measured incubation period of SARS-CoV-2 qRT-PCR measurements. Incubation period is defined as the time (hours) from inoculation to the first quantifiable of the two viral quantifiable positives used to assess infection, starting from 24 hours post-inoculation and up to discharge from quarantine.
Time Frame: From 24 hours post-inoculation until discharged from Quarantine, up to a maximum period of 16 days
Measure: Mean (Standard Deviation); unit: Incubation Period (Hours) (Mid-Turbinate
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Incubation Period (Hours) (Mid-Turbinate | 75.527 (35.8999)

12. Secondary Outcome: SARS-CoV-2 Induced Symptoms in Healthy Volunteers According to Area Under the Curve Over Time (TSS-AUC) of Total Clinical Symptoms (TSS).
Description: Area under the curve over time (TSS-AUC) of total clinical symptoms (TSS) as measured by graded symptom scoring system (categorical and visual analogue scales), starting one day post-viral challenge (Day 1) up to discharge from quarantine. Symptoms are graded on a scale from 0 (no symptoms) to 3 (bothersome symptoms impacting involvement in activities). The sum total symptom score was based on the symptom diary cards that were filled out 3 times per day from the first (morning) assessment on Day 1 until the first (morning) assessment on Day 14 (planned day of quarantine discharge). Each assessment consisted of the grades given by the subjects to a list of 19 symptoms on the symptom diary card. Individual total symptom scores were derived for each assessment as the total of all of the grades given on the individual diary card. This could range from 0 (if all symptoms graded as 0) to 59 (if all symptoms graded as 3 and shortness of breath and wheeze were graded as 4).
Time Frame: From 24 hours post-inoculation to 312 hours post-inoculation
Measure: Mean (Standard Deviation); unit: Total Symptom Score AUC (hours*score)
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Total Symptom Score AUC (hours*score) | 213.444 (337.8488)

13. Secondary Outcome: SARS-CoV-2 Induced Symptoms in Healthy Volunteers According to Peak Symptom Diary Card Scores
Description: Peak symptoms diary card score: peak total clinical symptoms (TSS) as measured by graded symptom scoring system (categorical and visual analogue scales, starting one day post-viral challenge (Day 1) up to discharge from quarantine. Symptoms are graded on a scale from 0 (no symptoms) to 3 (bothersome symptoms impacting involvement in activities). The sum total symptom score was based on the symptom diary cards that were filled out 3 times per day from the first (morning) assessment on Day 1 until the first (morning) assessment on Day 14 (planned day of quarantine discharge). Each assessment consisted of the grades given by the subjects to a list of 19 symptoms on the symptom diary card. Individual total symptom scores were derived for each assessment as the total of all of the grades given on the individual diary card. This could range from 0 (if all symptoms graded as 0) to 59 (if all symptoms graded as 3 and shortness of breath and wheeze were graded as 4).
Time Frame: From 24 hours post-inoculation until 312 hours post-inoculation
Measure: Mean (Standard Deviation); unit: Peak Total Symptom Score
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Peak Total Symptom Score | 2.8 (2.86)

14. Secondary Outcome: SARS-CoV-2 Induced Symptoms in Healthy Volunteers According to Peak Daily Symptom Score.
Description: Peak daily symptom score: Individual maximum daily sum of Symptom score starting one day post-viral challenge (Day 1) up to the end of quarantine. Symptoms are graded on a scale from 0 (no symptoms) to 3 (bothersome symptoms impacting involvement in activities). The sum total symptom score was based on the symptom diary cards that were filled out 3 times per day from the first (morning) assessment on Day 1 until the first (morning) assessment on Day 14 (planned day of quarantine discharge). Each assessment consisted of the grades given by the subjects to a list of 19 symptoms on the symptom diary card.
  Individual total symptom scores were derived for each assessment as the total of all of the grades given on the individual diary card. This could range from 0 (if all symptoms graded as 0) to 59 (if all symptoms graded as 3 and shortness of breath and wheeze were graded as 4).
Time Frame: From 24 hours post-inoculation until 312 hours post-inoculation
Measure: Mean (Standard Deviation); unit: Peak Daily Total Symptom Score
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Peak Daily Total Symptom Score | 5.8 (6.98)

15. Secondary Outcome: Number (%) of Participants With Grade 2 or Higher SARS-CoV-2 Induced Symptoms
Description: Number (%) of participants with Grade 2 or higher symptoms. Symptoms are graded on a scale from 0 (no symptoms) to 3 (bothersome symptoms impacting involvement in activities). The sum total symptom score was based on the symptom diary cards that were filled out 3 times per day from the first (morning) assessment on Day 1 until the first (morning) assessment on Day 14 (planned day of quarantine discharge). Each assessment consisted of the grades given by the subjects to a list of 19 symptoms on the symptom diary card. Individual total symptom scores were derived for each assessment as the total of all of the grades given on the individual diary card. This could range from 0 (if all symptoms graded as 0) to 59 (if all symptoms graded as 3 and shortness of breath and wheeze were graded as 4).
Time Frame: From 24 hours post-inoculation until 312 hours post-inoculation
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Participants | 14

16. Other Pre Specified Outcome: Average Change in Smell Measured by the University of Pennsylvania Smell Identification Test (UPSIT)
Description: To explore safety related measures of wild type SARS-CoV-2 challenge in healthy participants by assessing changes in smell (anosmia/parosmia) measured by the University of Pennsylvania Smell Identification Test (UPSIT). The USPIT test has 40 smells to "scratch and sniff". Each smell has a possible of 4 answers with one being correct, therefore the potential scores can range from 0-40.
  Score of less than 19 = anosmia. Score of 19 to 25 = severe microsmia. Score of 26 to 30 in females or 26 to 29 in males = microsmia Score of 31 to 24 in females or 30 to 33 in males = mild microsmia Score of 35 or more in females or 34 or more in males = normosmia
Time Frame: Day 0 to 28 (28 days)
Measure: Mean (1% Confidence Interval); unit: score on a scale
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
score on a scale | -0.5 [-0.5 to -0.5]

17. Other Pre Specified Outcome: Average Pulmonary Changes Measured by Spirometry (FEV1, FVC)
Description: To explore the safety of wild type SARS-CoV-2 human challenge model in healthy adults by assessing pulmonary changes due to experimental infection, as measured by Spirometry FEV1 and FVC. FEV1 and FVC will both be used for FEV1/FVC ratio.
Time Frame: Day 0 to 28 (28 days)
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Healthy Volunteers: Healthy volunteers given SARS-CoV-2 virus +/- Remdesivir: VEKLURY™
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 36
ratio | -0.4 (4.06)

18. Other Pre Specified Outcome: Number of Haematological and Biochemical Laboratory Abnormalities During the Quarantine Period
Description: To explore the safety of wild type SARS-CoV-2 human challenge model in healthy adults by assessing the occurrence of haematological and biochemical laboratory abnormalities during the quarantine period. Haematological and biochemical laboratory abnormalities will be identified from blood sampling analysis.
Time Frame: Day 0 to 28 (28 days)
Measure: Number; unit: Laboratory Test Results reported as AEs
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Laboratory Test Results reported as AEs | 13

19. Other Pre Specified Outcome: Number of Participants Using Concomitant Medication Within 30 Days Post-viral Challenge
Description: To explore the safety of wild type SARS-CoV-2 human challenge model in healthy adults by assessing the use of concomitant medications within 30 days post-viral challenge (Day 0 up to Day 28 follow up).
Time Frame: Day 0 to 28 (28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Volunteers Dose Level 1
Number analyzed (Participants) | 36
Participants | 26

ADVERSE EVENTS:
Time Frame: Day 0 to Day 360
Arm/Group | Healthy Volunteers Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 24/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers Dose Level 1 (N=36)
Left Side Renal Pain (Renal and urinary disorders) | 1 (1) — One participant experienced severe left side renal pain from 10 Dec 2021 to 31 Dec 2021 (Day 183 to Day 204). This was classed as not related to viral challenge and possibly related to passing of renal calculi. The subject was hospitalised.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteers Dose Level 1 (N=36)
Fibrin D dimer increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Troponin increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Medical device site rash (General disorders) | 5
Vessel puncture site bruise (General disorders) | 1
Catheter site rash (General disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Anosmia (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
COVID-19 (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Epididymal tenderness (Reproductive system and breast disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04865237/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT04865237/SAP_001.pdf